CLINICAL TRIAL: NCT06723483
Title: Results of Usage of Bridging Plate in Multi-fragmentary Distal Radius Fracture
Status: Active, not recruiting | Type: Observational
Sponsor: Mina Hany Moris Zakhary (Other)
Responsible Party: Sponsor-Investigator, Mina Hany Moris Zakhary, Resident doctor, Assiut University
Organization: Assiut University (Other)
Other Study IDs: 04-2024-200841
Record Dates: First submitted 2024-10-03; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Distal Radius Fractures; Mechanical Complication of Internal Rod Fixation Device; Internal Fixation; Complications
Keywords: bridging plate, distraction plate
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Distraction Plate — This technique deals with comminuted distal radius fracture using a distraction plate. The plate was inserted by minimally invasive skin incisions, fixed from the 2end metacarpal distally to the 2end extensor compartment at intact radius proximally Spaning the comminution, Restoring the Radial Length, Radial Inclination, Volar Tilt
  Other Names: bride plating; bridging plate

SUMMARY:
using a plate as a distraction method bridging the comminution to restore anatomical parameters to treat comminuted distal radius fracture follow-up functional outcomes of the wrist after metal removal

DETAILED DESCRIPTION:
The plate is extended from the floor of the 2end extensor compartment at an intact radius to the 2end metacarpal by dual minimally invasive skin incisions.

One distal over 2end metacarpal and Other proximal over 2end extensor compartment at intact radius application of distal screws 1st, then the traction is done to restore radial length, radial inclination, and volar tilt followed by the application of proximal screws add wires to restore the joint congruity wire removal after 45 days, plate removal after 100 day follow up every 3 months till 1 year post-operative Assess the Functional Outcome Of the wrist joint after metal removal

ELIGIBILITY:
Inclusion Criteria:

1. Skeletally mature patients
2. presented with multifragmentary distal radius fractures classify type 23-3C according to AO classification
3. articular with or without metaphyseal comminution
4. Very distal fractures 5 )osteoporotic bone fractures

Exclusion Criteria:

1. Dorsal soft tissue defect or tendon injuries
2. Metacarpal fractures (esp 2end MC)
3. open grade 3 fractures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: oFirst peak is the young exposed to high energy trauma , fall from a height, polytrauma patients with extensive communition of metaphyseal and articular parts oSecond peak is old (over 60 years),with osteoporotic bone where even minor falls can cause extensive comminution
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Modified Mayo Wrist Score (MMWS) | Mean follow-up period is 1 year postoperative.
  Combines subjective and objective parameters to evaluate wrist functionality.

SECONDARY OUTCOMES:
Wrist Range of Movement | Mean follow-up period is 1 year postoperative.
  Measurements include:
  Flexion (degrees) Extension (degrees) Pronation (degrees) Supination (degrees) Each measurement will be assessed separately using a goniometer.

CONTACTS AND LOCATIONS:
Overall Officials: Waleed Riad Saleh Waleed Riad Saleh Ramadan, preso doctor, Study Chair — assiut university hospitals; Yasser Farouk Yasser Mohamed Farouk Fouad Ragheb, doctor, Study Director — assiut university hospitals
Locations (1):
- Faculty of medicine assuit university, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Yes